CLINICAL TRIAL: NCT03170557
Title: A Randomized, Double Blind, Comparative Trial to Assess the Efficacy of Traditional Acupuncture vs Aspecific Needle Skin Stimulation for Persistent Pain in Subjects With Spinal Cord Injury
Brief Title: Randomized Comparative Trial for Persistent Pain in Spinal Cord Injury: Acupuncture vs Aspecific Needle Skin Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After a first stop due to acupuncturists unavailability, the Covid-19 pandemic also impacted on the study time schedule for acupuncture administration and outcomes evaluation.
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Collaborators: Associazione Medici Agopuntori Bolognesi (A.M.A.B.) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-17017
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pain; Spinal Cord Injuries
Keywords: Persistent pain; Spinal cord injury; Acupuncture; Randomized Controlled Trial; RCT
MeSH Terms: conditions — Pain; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized comparative trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician in charge for data analysis will be blind with respect to the identity of the assignment Groups (that will be coded so as not to be recognized) and will not be involved in filling data in the database to be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional chinese acupuncture (Active Comparator): Traditional chinese acupuncture. Administration of 12 sessions (2 per week for 6 weeks). Each session lasts 20-30 minutes.
  Interventions: Other: Traditional chinese acupuncture
- Aspecific needle skin stimulation (Sham Comparator): Aspecific needle skin stimulation. Administration of 12 sessions (2 per week for 6 weeks). Each session lasts 20-30 minutes.
  Interventions: Other: Aspecific needle skin stimulation

INTERVENTIONS:
Other: Traditional chinese acupuncture — Traditional chinese acupuncture (somatopuncture points, auriculotherapy points, craniopuncture and wrist-ankle acupuncture). Simultaneously, the usual pharmacological treatment for pain is maintained, based on clinical needs.
  Arms: Traditional chinese acupuncture
Other: Aspecific needle skin stimulation — Superficial needling of needles in skin areas outside the pain affected dermatome(s). Simultaneously, the usual pharmacological treatment for pain is maintained, based on clinical needs.
  Arms: Aspecific needle skin stimulation

SUMMARY:
Pain is one of the most common problems in patients with spinal cord injury (SCI) and persistent pain (that can be of different origin: nociceptive, neuropathic or mixed) is often poorly responsive to pharmacological therapy. Attention has been paid to the use of non-pharmacological therapies and interventional techniques in treating pain in other clinical conditions, and acupuncture has been the treatment most used and appreciated for its effectiveness. However, only few studies are available on the use of acupuncture in SCI patients. The present randomized, comparative trial aims to clarify the efficacy of traditional acupuncture vs. aspecific needle skin stimulation in treating persistent pain in subjects with spinal cord injury, by overcoming the biases reported in previous studies.

DETAILED DESCRIPTION:
About 67% of patients with spinal cord injury (SCI) experience painful symptoms in the course of life after injury and a third evaluates the pain as "severe", with a significant impact on quality of life, due to limitations in daily activities and autonomy. Persistent pain can be of different origin and may be nociceptive, neuropathic or mixed. However, it is often poorly responsive to pharmacological therapy. For some years, attention has been paid to the use of non-pharmacological therapies and interventional techniques in treating pain, and acupuncture has been the treatment most used and appreciated for its effectiveness. Only two studies on the use of acupuncture in SCI patients were included in the only Cochrane review available, dated 2014. Such studies, focusing on the painful shoulder syndrome and, therefore, on skeletal muscle pain, show a "non-superiority" of acupuncture compared to sham acupuncture treatment or Trager approach. However, the review does not come to any clear conclusions on the effectiveness of intervention because of the small number of cases and high risk of bias.

A more recent primary, randomized, controlled trial on SCI patients, although focusing on chronic pain and on a single acupuncture technique, uses a questionable study design (cross-over) to demonstrate treatment efficacy.

The present randomized, comparative trial aims to clarify the efficacy of traditional acupuncture vs. aspecific needle skin stimulation in treating persistent pain in subjects with spinal cord injury, by overcoming the biases reported in previous studies. Because of the intrinsic effects of sham acupuncture and, generally, of skin stimulation, a statistically significant change in the Numerical Rating Scale (NRS) measurements is expected even in the comparison group. To minimize this bias, which cannot be avoided, and to maintain the blindness of the patient as much as possible, the comparison group is treated by the insertion of needles in skin areas outside the metamer(s) affected by pain.

Primary objective:

- To evaluate the efficacy of traditional acupuncture vs. aspecific needle skin stimulation for persistent pain in subjects with spinal cord injury, at the end of treatment and at the 3 week follow-up.

Secondary objectives:

* Reduction of drug intake, at the end of treatment and at the subsequent follow-up;
* Reduction of anxiety/depression, at the end of treatment and at the subsequent follow-up;
* Improvement of quality of life, at the end of treatment and at the subsequent follow-up;
* Persistence of the effect of acupuncture 9 weeks after treatment.

Data concerning any adverse events, related to both experimental treatments of the trial, will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Persistent pain: NRS score >2 in at least 5 assessments in 5 consecutive days, despite usual antalgic management;
* Spinal cord injury due to any etiology (both traumatic and non-traumatic);
* Spinal cord injury of any neurological level, complete or incomplete, classifiable as Asia Impairment Score (AIS) A, B, C or D;
* Stable medical conditions;
* At least 1 month away from the spinal cord injury event.

Exclusion Criteria:

* Sporadic pain;
* Mechanical ventilation;
* Pregnancy;
* Disorders of consciousness;
* Incapacity to give informed consent in person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Pain reduction | Baseline (initial visit); session 6 (3 weeks); closing session 12 (6 weeks); follow-up 1 (3 weeks after closing session 12)
  Pain reduction of at least 2 points on the NRS scale

SECONDARY OUTCOMES:
Persistence of pain reduction in Acupuncture arm | Follow-up 2 (9 weeks after closing session 12)
  Pain reduction of at least 2 points on the NRS scale
Reduction of drugs intake | Baseline (initial visit); session 6 (3 weeks); closing session 12 (6 weeks); follow-up 1 (3 weeks after closing session 12); follow-up 2 (9 weeks after closing session 12)
  Intake reduction of antalgic, hypnotic and anxiolytic drugs (number and dosage)
Reduction of Anxiety/Depression | Baseline (initial visit); closing session 12 (6 weeks); follow-up 1 (3 weeks after closing session 12); follow-up 2 (9 weeks after closing session 12)
  Reduction of anxiety/depression symptoms, assessed by Hospital Anxiety and Depression Scale
Reduction of pain interference on sleep and quality of life | Baseline (initial visit); closing session 12 (6 weeks); follow-up 1 (3 weeks after closing session 12)
  Reduction of pain interference on sleep and quality of life, assessed by Multidimensional Pain Inventory scale, Part 1
Improvement of quality of life | Baseline (initial visit); closing session 12 (6 weeks); follow-up 2 (9 weeks after closing session 12)
  Increase of participation in family and social life, assessed by Multidimensional Pain Inventory scale, Part 2

OTHER OUTCOMES:
Patient satisfaction | Closing session 12 (6 weeks)
  Assessment of patient satisfaction after antalgic treatment by an in-house developed ad-hoc questionnaire
Adverse events | Session 6 (3 weeks); closing session 12 (6 weeks); follow-up 1 (3 weeks after closing session 12)
  Recording possible adverse events attributable to the experimental treatments

CONTACTS AND LOCATIONS:
Overall Officials: Angela Morreale, MD, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided